CLINICAL TRIAL: NCT06860490
Title: Sintilimab Plus Bevacizumab Biosimilar with or Without HAIC for Advanced Hepatocellular Carcinoma (TASK-03): a Multicenter, Randomized, Phase 2 Study
Brief Title: HAIC Combined with Sintilimab Plus Bevacizumab Biosimilar for Advanced Hepatocellular Carcinoma (TASK-03)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASK-03
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAIC+sintilimab+bevacizumab (Experimental): HAIC in combination with Sintilimab plus bevacizumab biosimilar
  Interventions: Drug: Sintilimab; Drug: Bevacizumab Biosimilar; Procedure: HAIC
- Sintilimab+bevacizumab (Active Comparator): Sintilimab plus bevacizumab biosimilar
  Interventions: Drug: Sintilimab; Drug: Bevacizumab Biosimilar

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be administered by IV, 200 mg on day 1 of each 21 day cycle.
Drug: Bevacizumab Biosimilar — Bevacizumab biosimilar will be administered by IV, 15 mg/kg on day 1 of each 21 day cycle.
Procedure: HAIC — FOLFOX regimen (oxaliplatin, 85 mg/m2 from hour 0-2 on day 1; leucovorin, 400 mg/m2 from hour 2-3 on day 1; and ﬂuorouracil, 400 mg/m2 bolus at hour 3 on day 1 and 2,400 mg/m2 over 24 hours) via infusion via the hepatic artery. HAIC was repeated once every 3 weeks for up to four cycles. Sintilimab plus bevacizumab will be administered 1-3 days after HAIC.
  Arms: HAIC+sintilimab+bevacizumab

SUMMARY:
To evaluate HAIC combined with Sintilimab plus bevacizumab biosimilar for advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is a randomized, multicenter, phase II study to determine the efficacy and safety of Sintilimab plus bevacizumab biosimilar combined with hepatic arterial infusion chemotherapy (HAIC) compared to Sintilimab plus bevacizumab biosimilar in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Barcelona Clinic Liver Cancer stage C, or stage B not amenable to curative or locoregional therapies.
* HCC conﬁrmed by radiology, histology or cytology.
* No prior systemic therapy for HCC.
* At least one measurable site of disease as defined by RECIST1.1criteria with spiral CT scan or MRI.
* Child-Pugh scores 5-7, performance status (PS) ≤ 2 (ECOG scale).
* Subjects with chronic HBV infection must have HBV DNA viral load < 100 IU/mL at screening. In addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy.
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥60 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula)
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* Patients on a liver transplantation list or with advanced liver disease.
* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Prior systemic anti-cancer therapy OR endocrine- OR immunotherapy.
* Prior treatment with HAIC.
* Radiotherapy administered less than 4 weeks prior to study treatment start.
* Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Previous treatment in the present study (does not include screening failure).
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to: a) history of interstitial lung disease b) Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection) c) known acute or chronic pancreatitis d) active tuberculosis e) any other active infection (viral, fungal or bacterial) requiring systemic therapy f) history of allogeneic tissue/solid organ transplant g) diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment. h) Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study. i) Live vaccine within 30 days prior to the first dose of treatment or during study treatment. j) History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS.
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2028-03-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  PFS is defined as the time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by investigator.
Disease control rate (DCR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD)
Duration of Response (DOR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DOR is defined as the time from first documented complete or partial response until disease progression, death from any cause, or censoring at date of last tumor assessment.
Time to Response (TTR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  TTR is defined as the time from the start of treatment until the first objective observation of a response (either partial response, PR, or complete response, CR), provided that the response is subsequently confirmed
Overall survival (OS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 42 months
  OS is defined as the time from study treatment to the date of death of the subject, regardless of the cause of death
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | max 42 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported
Translational study | max 42 months
  Proportion of different immune cell types in tumors based on single-cell RNA sequencing between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided